CLINICAL TRIAL: NCT00861835
Title: A Randomized Prospective Trial of Rapid On-Site Evaluation of Transbronchial Needle Aspirate Specimens
Brief Title: Trial of Rapid On-Site Evaluation of Transbronchial Needle Aspirate (TBNA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Lonny Yarmus, DO, Maine Medical Center
Purpose: Diagnostic
Other Study IDs: MMCROSE
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ROSE for TBNA (Experimental)
  Interventions: Other: ROSE
- NR (No Intervention): no on-site cytopathology assessment (NR)

INTERVENTIONS:
Other: ROSE — rapid on-site evaluation by cytopathology
  Arms: ROSE for TBNA

SUMMARY:
Purpose: Previous studies suggested an increased diagnostic yield for bronchoscopic (FB) transbronchial needle aspirate (TBNA) specimens from mediastinal lymph nodes when using rapid on-site evaluation by cytopathology (ROSE) but were limited by lack of randomization. The investigators performed the first randomized-prospective trial comparing ROSE(R) to no on-site cytopathology assessment (NR).

Methods: All patients referred were eligible. 78 patients were randomized to R or NR groups. For R procedures, further specimens were deferred until results were available from the on-site cytopathologist. Diagnoses made by all procedures were recorded. The primary end-points were specimen adequacy and diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients included all adults referred for bronchoscopy with anticipated TBNA.

Exclusion Criteria:

* Patients were to be excluded only if the attending physician felt ROSE must be used for diagnosis or if the patient refused consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
diagnostic yield